CLINICAL TRIAL: NCT05365178
Title: A Randomized, Double-blind, Parallel-controlled Phase III Trial Evaluating the Efficacy and Safety of TQB3616 in Combination With Fulvestrant Versus Placebo in Combination With Fulvestrant in Previously Untreated HR-positive, HER2-negative Advanced Breast Cancer
Brief Title: To Evaluate the Efficacy and Safety of TQB3616 in Combination With Fulvestrant Versus Placebo in Combination With Fulvestrant in Previously Untreated Hormone-receptor (HR)-Positive, Human Epidermal Growth Factor Receptor 2 (HER2)-Negative Advanced Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQB3616-Ⅲ-02
Record Dates: First submitted 2022-04-26; First posted 2022-05-09 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-07

CONDITIONS: HR-positive, HER2-negative Breast Neoplasms
MeSH Terms: interventions — Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB3616 capsule + Fulvestrant injection (Experimental): TQB3616 capsule:
  180mg was given orally with meals or within 2 hours after meals, once a day， every 28 days for a cycle.
  Fulvestrant injection:
  500mg intramuscular injection was administered on day 1, every 28 days for a cycle, for the first cycle, was administered on day 1 and day 15
  Interventions: Drug: TQB3616 capsule; Drug: Fulvestrant injection
- Placebo capsule + Fulvestrant injection (Placebo Comparator): Placebo capsules:
  0mg was given orally with meals or within 2 hours after meals, once a day, every 28 days for a cycle.
  Fulvestrant injection:
  500mg intramuscular injection was administered on day 1, every 28 days for a cycle, for the first cycle, was administered on day 1 and day 15
  Interventions: Drug: Placebo; Drug: Fulvestrant injection

INTERVENTIONS:
Drug: TQB3616 capsule — TQB3616 capsule is a CDK (cyclin-dependent kinases) 2/4/6 kinase inhibitor, which can selectively inhibit THE activity of CDK2/4/6 kinase, make it form a complex with Cyclin D, reduce the phosphorylation level of retinoblastoma protein (Rb) in cancer cells, and prevent cells from entering S phase from G1 phase
  Arms: TQB3616 capsule + Fulvestrant injection
Drug: Placebo — It is a placebo
  Arms: Placebo capsule + Fulvestrant injection
Drug: Fulvestrant injection — Fulvestrant is a competitive estrogen receptor antagonist, and its mechanism is related to the down-regulation of estrogen receptor (ER) protein level

SUMMARY:
A randomized, double-blind, parallel-controlled, multicenter trial design was used in this study. Subjects who meet the criteria will be randomly divided into 2:1 groups to receive TBQ3616 capsule combined with Fulvestrant injection (experimental group) or placebo capsule combined with fulvestrant (control group). A total of 428 subjects were required.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in this study and sign informed consent with good compliance;
* Age: 18-75 years (when signing the informed consent); an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1; Is expected to survive more than 3 months;
* Postmenopausal or premenopausal/perimenopausal women；
* Patients with HR-positive or HER2-negative breast cancer confirmed by pathological examination with evidence of local lesion recurrence or distant metastasis, not suitable for the surgery or radiotherapy for the purpose of cure, and there are no clinical indications of chemotherapy；
* Have a measurable lesion (RECIST (Response Evaluation Criteria In Solid Tumors) 1.1 criteria), or have only bone metastases；
* The main organs function well and meet the following standards：

  1. Routine blood examination should meet the following criteria: (No blood transfusion and no hematopoietic stimulation drugs within 7 days before screening)

     1. Hemoglobin (HB) ≥100 g/L;
     2. Absolute value of neutrophils (NEUT) ≥ 1.5×109/L;
     3. Platelet count (PLT) ≥ 90 ×109/L.
  2. Biochemical blood tests shall meet the following criteria：

     1. Total bilirubin (TBIL) ≤ 1.5 times normal upper limit (ULN);
     2. Alanine transferase (ALT) and aspartate transferase (AST) ≤ 2.5×ULN; ALT and AST≤ 3×ULN for patients with liver metastasis;
     3. Serum creatinine (Cr) ≤ 1.5×ULN, or creatinine clearance (Ccr) ≥ 60 mL /min；
  3. Coagulation function tests shall meet the following criteria：

     (a) Prothrombin time (PT), activated partial thrombin time (APTT), international standardized
  4. Color doppler echocardiography: Left ventricular ejection fraction (LVEF) ≥50%；
* Female subjects within reproductive age should agree to use contraceptive methods (such as intrauterine devices, birth control pills or condoms) from participating the study to 6 months after the end of the study; Serum pregnancy test result should be negative within 7 days prior to study enrollment and must be non-lactating subjects.

Exclusion Criteria:

* Associated diseases and history：

  1. The presence or current co-occurrence of other malignant tumors within 5 years, except ured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor infiltrating basal membrane)];
  2. Multiple factors affecting oral and drug absorption (such as inability to swallow, post-gastrointestinal resection, ulcerative colitis, symptomatic/inflammatory bowel disease, chronic diarrhea and intestinal obstruction);
  3. Patients with a history of severe pneumonia such as interstitial lung disease;
  4. Unrelieved toxicity higher than GRADE 1 Common Terminology Criteria for Adverse Events (CTCAE) due to any previous anti-tumor treatment, hair loss is not included;
  5. Major surgery or significant traumatic injury within 28 days prior to randomization;
  6. Long-term unhealed wounds, ulcers or fractures;
  7. Occurrence of arteriovenous/venous thrombosis events within 6 months, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc.;
  8. History of psychotropic drug abuse and can't get rid of it or with mental disorders;
  9. Subject with any severe and/or uncontrolled disease, including：

     1. Arrhythmias requiring treatment with grade≥2 myocardial ischemia, myocardial infarction, and congestive heart failure (NYHA(New York Heart Association) classification) within 6 months prior to study enrollment (including qtc≥480ms during screening period); And uncontrolled high blood pressure;
     2. Active or uncontrolled severe infection (≥CTCAE grade 2 infection) or unexplained fever > 38.5℃ within 28 days prior to randomization;
     3. Decompensated cirrhosis (Child-Pugh liver function score B or C), active hepatitis ;
     4. Patients with renal failure requiring hemodialysis or peritoneal dialysis;
     5. A history of immunodeficiency, including HIV ( Human Immunodeficiency Virus) positive or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation or hematopoietic stem cell transplantation;
* Tumor-related symptoms and treatment；

  1. Visceral crisis exists;
  2. Severe bone injury due to bone metastasis of tumor;
  3. Received radiotherapy (except palliative radiotherapy for non-target lesions) and other anti-tumor therapies (the washout period was calculated from the end of the last treatment) within 2 weeks prior to randomization;
  4. Prior medical treatment with fulvestrant, everolimus or CDK4/6 inhibitor;
  5. The presence of clinically uncontrolled pleural, ascites and pericardial effusion requiring repeated drainage or medical intervention (14 days prior to randomization);
* Known allergy to fulvestrant, Luteal Hormone Releasing Hormone (LHRH) agonists (e.g. Goserelin), TQB3616/ placebo or any supplement;
* History of live attenuated vaccine vaccination within 28 days prior to randomization or planned live attenuated vaccine vaccination during the study period;
* Participated in clinical trials of other antitumor drugs within 4 weeks pior to randomization;
* With other serious physical or mental diseases or abnormal laboratory tests that may increase the risk of study participation or interfere with the study results, or unsuitable for the study for other reasons considered by investigators.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival as assessed by the investigator | Baseline up to progressive disease (PD)/die, about 25.8 months
  The time from enrollment to the date of the first documentation of objective progression of disease or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression-free survival (PFS) by independent imaging assessment | Baseline up to PD/die, about 25.8 months
  The time from enrollment to the date of the first documentation of objective progression of disease or death due to any cause, whichever occurs first.
Overall survival | Baseline up to die, about 36months
  Overall survival was defined as the time from randomization to death from any cause.
3-Year Overall Survival (OS) | Baseline to 3 years
  The percentage of participants of survival above 3 years
Objective Response Rate (ORR) | Baseline to CR/PR，about 1 year
Clinical Benefit Rate(CBR) | Baseline to CR/PR/SD，about 1 year
  Calculated as the percentage of participants with best overall response of CR, PR, stable disease (SD) and Non-CR/Non-progressive disease (PD).
Duration of Overall Response (DOR) | CR/PR assessment, up to PD/die, about 20 months
  The time from the date of participants with a first overall response defined as complete response (CR) or partial response (PR) to the date of the first documentation of objective progression of disease or death due to any cause, whichever occurs first.
The European Organization for Research and Treatment of Cancer Quality of Life questionnaire | Baseline to the end of the study, about 3 years
  Sense of satisfaction, life quality of participants since the enrollment of the study
Incidence of adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs). | Baseline to the end of the study, about 3 years
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).

CONTACTS AND LOCATIONS:
Locations (88):
- China (88):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - The Southwest Hospital of AMU, Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Gansu Wuwei Tumour Hospital, Wuwei, Gansu
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Nanfang Hospital Southern Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Jieyang People's Hospital, Jieyang, Guangdong
  - Maoming people's hospital, Maoming, Guangdong
  - Yue Bei People's Hospital, Shaoguan, Guangdong
  - ShenZhen People's Hospital, Shenzhen, Guangdong
  - PeKing University ShenZhen Hosipital, Shenzhen, Guangdong
  - Zhongshan City People's Hospital, Zhongshan, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat-Sen University, Zhuhai, Guangdong
  - The Second Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Yulin First People's Hospital, Yulin, Guangxi
  - The Affiliated Hospital of Hebei University, Baoding, Hebei
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Hebei Cangzhou Hospital of Integrated Traditional Chinese, Cangzhou, Hebei
  - Affiliated Hospital of Chengde Medical University, Chengde, Hebei
  - Hebei Petro China Central Hospital, Langfang, Hebei
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Affiliated Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Jiamusi Cancer Hospital, Jiamusi, Heilongjiang
  - Luoyang Central Hospital, Luoyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Yichang Central People's Hospital, Yichang, Hubei
  - The First People's Hospital of Changde, Changde, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Changzhou Cancer Hospital, Changzhou, Jiangsu
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jiangsu province hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - The Third Hospital of Nanchang, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - Second Hospital of Jilin University, Changchun, Jilin
  - The Second Hosptial of DaLian Medical University, Dalian, Liaoning
  - Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Affiliated Hospital of Chifeng University, Chifeng, Neimenggu
  - Inner Mongolia Autonomous Region Cancer Hospital, Hohhot, Neimenggu
  - The Affilliate Hospital of Inner Mongolia Medical Univercity, Hohhot, Neimenggu
  - General Hospital of Ningxia Medical, Yinchuan, Ningxia
  - Qinghai University affiliated hospital, Xining, Qinghai
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - First Affiliated University Hospital of PLA Air Force Military Medical, Xi'an, Shaanxi
  - Second Affiliated Hospital of PLA Air Force Military Medical, Xi'an, Shaanxi
  - Xi'an International Medical Center Hospital, Xi'an, Shaanxi
  - Binzhou Medical College Affiliated Hospital, Binzhou, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Linyin Cancer Hospital, Linyi, Shandong
  - Qingdao University Affiliated Hospital, Qingdao, Shandong
  - Weifang Hospital of Traditional Chinese Midicine, Weifang, Shandong
  - Yantai Yantai Mountain hospital, Yantai, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - Huadong Hospital, Shanghai, Shanghai Municipality
  - Shanghai Oriental Hospital, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - Changzhi People's Hospital, Changzhi, Shanxi
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Chinese People's Liberation Army Western Theater General Hospital, Chengdu, Sichuan
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Hospital Konggang Hospital, Tianjin, Tianjin Municipality
  - Cancer Hospital affiliated to Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Cancel Hospital, Kunming, Yunan
  - Affiliated Hangzhou First People's Hospital, Zhejiang University School of Medcine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Xu Z, Liu Y, Song B, Ren B, Xu X, Lin R, Zhu X, Chen C, Yang S, Zhu Y, Jiang W, Li W, Xia Y, Hu L, Chen S, Chan CC, Li J, Zhang X, Yang L, Tian X, Ding CZ. Discovery and preclinical evaluations of TQB3616, a novel CDK4-biased inhibitor. Bioorg Med Chem Lett. 2024 Jul 15;107:129769. doi: 10.1016/j.bmcl.2024.129769. Epub 2024 Apr 24. PMID 38670537